CLINICAL TRIAL: NCT06511284
Title: Swallowing and Nutritional Therapy and Its Impact on Body Composition and Clinical Outcomes in Patients With Post-extubation Dysphagia
Brief Title: Nutritional Therapy in Patients With Post-extubation Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Ivan Armando Osuna Padilla, Clinical Nutrition Manager, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C32-24
Record Dates: First submitted 2024-07-10; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Dysphagia
Keywords: enteral nutrition; nutritional assessment; nutritional therapy; Deglutition Disorders; rehabilitation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Amounts of protein was not revealed for participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein group (Experimental): 100% of the energy requirements measured by indirect calorimetry (IC) or estimated, and a protein intake of 2.0 g/kg, will be prescribed
  Interventions: Other: High protein dose
- Usual protein group (Other): 100% of the energy requirements measured by IC or estimated, and a protein intake of 1.5 g/kg, will be prescribed.
  Interventions: Other: Usual protein dose

INTERVENTIONS:
Other: High protein dose — High dose of protein (2.0 g/kg) will prescribed for home enteral nutrition
  Arms: High protein group
Other: Usual protein dose — Usual dose of protein (1.5 g/kg) will prescribed for home enteral nutrition
  Arms: Usual protein group

SUMMARY:
The aim of this study is to evaluate the impact of the prescription of two doses of protein on the amount in kilograms of muscle mass and on the clinical evolution (time until safe swallowing, time until removal of the feeding stoma, number of hospital readmissions, feeding stoma infections, incidence of pneumonia, functionality, number of falls, fractures and mortality) at 6 months after hospital discharge in patients with enteral nutrition due to post-extubation dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required invasive mechanical ventilation during their hospital stay with a diagnosis of post-extubation dysphagia diagnosed by fibroendoscopy evaluation of swallowing (FEES).
* Patients who discharged with a feeding tube.
* Patients with signed informed consent.

Exclusion Criteria:

* Patients with pre-existing dysphagia, or with neurological conditions that can cause dysphagia (e.g. multiple sclerosis, Parkinson's disease, Alzheimer's, myasthenia gravis).
* Patients with chronic kidney disease, defined as a glomerular filtration rate <60 ml/min.
* Patients discharged with a terminal condition and/or life expectancy of less than 3 months.
* Diagnosis of HIV, upon receiving clinical follow-up by the team of specialists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass changes | From randomization to 6 months
  Changes of muscle mass in kilograms measured by impedance bioelectric

SECONDARY OUTCOMES:
Swallow recovery | From randomization to 6 months
  Time to safe swallowing diagnosed by fibroendoscopy evaluation of swallowing (FEES) and measured in months
Duration of enteral nutrition indication | From randomization to 6 months
  Time from discharge to feeding tube removal
Feeding tube complications | From randomization to 6 months
  Number of feeding tube infections, dysfunctions and oclusions during study period
Muscle functionality changes | From randomization to 6 months
  Changes in functionality measured by medical research council scale in a scale of 0-60 points
Handgrip strenght changes | From randomization to 6 months
  Changes in functionality assessed by handgrip strenght in kilogramos using a digital dynamometer
Frailty complications | From randomization to 6 months
  Number of falls and fractures during study period
Hospital readmissions associated to dysphagia complications | From randomization to 6 months
  Number of hospital readmissions assocciated to feeding tube infections, dysfunctions and oclusions during study period
6-month mortality | From randomization to 6 months
  All-cause mortality during study period
Aspiration pneumonia incidence | From randomization to 6 months
  Number of hospital readmissions due to aspiration pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Ivan A Osuna-Padilla, PhD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No